CLINICAL TRIAL: NCT00144430
Title: A Phase II Study of Pentostatin For the Treatment of High Risk or Refractory Chronic GVHD in Children
Brief Title: Pentostatin for High Risk and Refractory Chronic Graft Versus Host Disease in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: David Jacobsohn, MD, Children's Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GVH 0313; NCT00228826 (obsolete NCT alias)
Record Dates: First submitted 2005-08-31; First posted 2005-09-05 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Graft vs Host Disease
Keywords: chronic graft versus host disease; graft; host; transplant; stem cell; pediatric; GVH0313; leukemia
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome; Leukemia | interventions — Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pentostatin — The drug, Pentostatin, is given every 2 weeks. This drug will be given by intravenous (IV) infusion.

SUMMARY:
This is a multicenter trial through the Pediatric Blood and Marrow Transplant Consortium.

The Primary hypothesis of this study is that because of its effect as a potent immunosuppressive agent targeting lymphocytes, pentostatin will show a sustained response in pediatric subjects with severe chronic GVHD. Secondary hypotheses include that the infection and toxicity rate of pentostatin in this setting will be acceptable given its lack of severe myelosuppression, and subjects with refractory chronic GVHD will have significant QOL impairment and symptomatology. These may change as subjects are being treated for their chronic GVHD with pentostatin.

DETAILED DESCRIPTION:
To participate in this study, subjects must have diagnosed chronic Graft versus Host Disease that is refractory to therapy or that is considered high risk (i.e. low platelet count, progressive onset and greater than 50% of body surface area affected). Subjects must have not failed more than 2 immunosuppressive regimens in order to be considered for this trial. Eligible subjects will receive intravenous pentostatin every 2 weeks for 24 weeks. If the subject has had a complete response, the therapy will end at 24 weeks. If the subject has had a partial or mixed response or stable disease, they will continue on study receiving pentostatin for 52 weeks.

ELIGIBILITY:
Inclusion criteria:

* Allogeneic BMT or SCT recipients. Includes cord blood and peripheral blood.
* Age 0-21 years.

FOR REFRACTORY GROUP:

* Diagnosis of chronic GVHD, confirmed by biopsy of any organ after SCT. Given the variability among centers, biopsy needs to say, at the very least, "consistent with GVHD." If there is a medical contra-indication (such as severe sclerosis with poor wound healing) or the need for an open procedure to obtain a fascial biopsy then a photograph documenting the skin and abnormal ROM studies may be submitted instead. If current GVHD represents the same episode which was previously biopsied, then a new biopsy is not necessary. If the previous biopsy was for an episode that went into remission and this is a new episode of GVHD, then a new biopsy is necessary.

To be eligible for this portion of the study, a patient's chronic GVHD can be extensive or limited, as defined below:

* All subjects with extensive chronic GVHD are eligible. These subjects must meet the following criteria:

  * Generalized skin involvement (>50% BSA)
  * OR Localized skin involvement and/or liver dysfunction plus at least one of the following:

    * Liver histology showing chronic aggressive hepatitis, bridging necrosis, cirrhosis, or ductopenia.
    * Eye involvement (Schirmer's test with < 5 mm wetting)
    * Involvement of minor salivary glands or oral mucosa on lip biopsy
    * Involvement of any other target organs
  * OR Involvement of at least 2 target organs.(Target organs are listed below under "Examples of characteristic manifestations)
* Subjects with limited chronic GVHD (defined as those with skin involvement in less than 50% BSA or isolated organ involvement 51 are also eligible. Examples of these subjects would be those with limited sclerodermatous or fascial skin disease or oral disease that is unresponsive to therapy and may be debilitating to the patient. Subjects with isolated refractory liver chronic GVHD may go on study provided they have liver histology as above.

Examples of characteristic manifestations include:

* skin changes - rash, lichenoid changes, sclerodermatous changes, hypopigmentation, hyperpigmentation, loss of appendages (hair follicles, sweat glands), alopecia
* oral changes - erythema, lichenoid changes, ulceration
* hepatic involvement - obstructive jaundice, chronic hepatitis, cirrhosis
* GI involvement - nausea, vomiting, weight loss, esophageal dysmotility, malabsorption, chronic diarrhea, abdominal cramps
* sicca syndrome - dry eyes and mouth (decreased tearing, keratoconjunctivitis, oral mucosal erythema and ulcerations)
* other inflammatory conditions - myositis, arthritis, polyserositis

To be eligible for this portion of the study subjects must have refractory disease defined below:

* Development of new sites of disease while being treated for chronic GVHD* (These criteria can be met at any time post-transplant after treatment for chronic GVHD has begun. This includes subjects who develop new sites of disease while on steroid therapy, tapering steroid therapy, or other therapy. The only necessary elements are TREATMENT of chronic GVHD and NEW area of disease. -OR-
* Progression of an initially affected site of chronic GVHD while being treated for chronic GVHD, the chronic GVHD worsens. This type of patient has worsening of any initially affected area at any time. This includes subjects that are judged to be steroid-dependent, and once a taper of steroids is initiated, they flare in the same organ. -OR-
* Failure to improve despite at least 1 month of standard therapy (These subjects have shown no response (not improved but not worse) to cGVHD therapy. These therapies include, but are not limited to:

  * Prednisone at an average of 0.5 mg/kg/day or equivalent steroid.
  * Another immunosuppressive regimen (e.g.. FK506/MMF or photopheresis).

FOR HIGH-RISK GROUP:

* The vast majority of these subjects will be identified at initial diagnosis of chronic GVHD and will be subjects progressing from acute to chronic. These subjects are likely to be on steroids for acute GVHD and have skin changes that are rapidly shifting from simple erythema to a lichenoid/pebbly appearance consistent with chronic GVHD. For inclusion into this arm, the following are required:

  * Extensive skin involvement (>50%BSA) with either lichenoid or sclerodermatous changes.
  * Either one or both of the following high-risk features:

    * Thrombocytopenia (PLT<100,000)
    * Progressive onset ( i.e. Changes suggestive of progression from acute to chronic). This includes, but is not limited to, skin becoming increasingly scaly, pebbly, raised, and lymphedematous. It is not unusual to see this transition even before day 100, especially in non-myeloablative SCT and DLI. If there are any questions regarding these changes and whether they qualify, call the PI, Dr. David Jacobsohn, 773-880-3694.
  * A biopsy after SCT showing acute or chronic GVHD. A biopsy showing acute GVHD is acceptable if the clinical picture is progressing to chronic GVHD.
  * Patient is on prednisone ≥2 mg/kg/day (or equivalent dose if on another steroid) and has received more than 7 days of therapy.

Exclusion Criteria:

* More than two previous regimens to treat chronic GVHD. A regimen for the purpose of this study is defined as an adequate trial of an immunosuppressive or immunosuppressive combination (patient was given drug or drugs for 3 months unless there was clear progression during regimen).
* Calculated Cr. Clearance<30 ml/min/1.73m2
* Active infection not responding to oral or IV antibiotics.
* Subjects and families unwilling to firmly commit to return for follow-up doses and appointments.
* Use of any investigational agent in the past 30 days (this does not include the use of licensed agents for indications not listed in the package insert).
* Pregnancy or nursing mother; Females of child-bearing potential and sexually active males should use effective contraception while on study.
* Active veno-occlusive disease of the liver.
* Bronchiolitis obliterans (defined for the purpose of this study by respiratory symptoms such as shortness of breath or cough and FEV1<50%).
* Karnofsky performance score less than 40 (or Lansky performance less than 40 in subjects under 16 years of age).

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To estimate the response rate (CR and PR) of pentostatin when used to treat refractory-chronic GVHD in children. | To end of study

SECONDARY OUTCOMES:
To gather initial efficacy and safety data in high-risk untreated chronic GVHD in children. | To end of study
To evaluate toxicities of pentostatin when used to treat chronic GVHD in children. | To end of study
To evaluate quality of life (QOL) and symptoms at diagnosis and after therapy with pentostatin in pediatric patients with refractory chronic GVHD. | To end of study

CONTACTS AND LOCATIONS:
Overall Officials: David Jacobsohn, MD, MSc, Principal Investigator — Children's Memorial Hospital, Chicago, IL
Locations (25):
- United States (25):
  - Loma Linda University Medical Center, Loma Linda, California
  - Pediatric Medical Center for Northern California, Oakland, California
  - Nemour's Children's Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - All Children's Health System, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - LSUHSC, New Orleans, Louisiana
  - John's Hopkins, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia Presbyterian Medical Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Rainbow Babies and Children's, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Victor Aquino, MD, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Southwest Texas Methodist Hospital, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Jacobsohn DA, Gilman AL, Rademaker A, Browning B, Grimley M, Lehmann L, Nemecek ER, Thormann K, Schultz KR, Vogelsang GB. Evaluation of pentostatin in corticosteroid-refractory chronic graft-versus-host disease in children: a Pediatric Blood and Marrow Transplant Consortium study. Blood. 2009 Nov 12;114(20):4354-60. doi: 10.1182/blood-2009-05-224840. Epub 2009 Sep 10. PMID 19745067